CLINICAL TRIAL: NCT00308022
Title: A Prospective Randomized Controlled Trial Comparing High Frequency Percussive Ventilation With Conventional Mechanical Ventilation Utilizing Protective Lung Strategies in Patients With Acute Lung Injury/Acute Respiratory Distress Syndrome
Brief Title: Comparison Study of High Frequency Percussive Ventilation With Conventional Ventilation
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The PI is no longer with the University
Sponsor: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTSW IRB 022005-052
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Distress Syndrome, Adult; Pneumonia; Mechanical Ventilation
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; High Frequency Percussive Ventilation; Ventilator Associated Pneumonia
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia; Acute Lung Injury; Pneumonia, Ventilator-Associated

INTERVENTIONS:
Device: High Frequency Percussive Ventilation

SUMMARY:
This study is designed to exam the effects of early management with high frequency percussive ventilation (HFPV) on patients with lung injury. Patients at risk for Acute Respiratory Distress Syndrome (ARDS) will be enrolled and randomized to one of two groups. One group will be managed with HFPV. The second group will be managed with conventional ventilation utilizing lung protective techniques. The primary endpoint of the study is rate of ventilator associated pneumonia. We hypothesized that use of HFPV in patients at risk for the development of ARDS will decrease the rate of ventilator associated pneumonia when compared to patients managed with conventional ventilation.

DETAILED DESCRIPTION:
Specific Aim 1: This prospective randomized trial will enroll 180 patients with ALI/ARDS over a forty-eight month period. One cohort will receive conventional mechanical ventilation adhering to our well defined protocol of protective lung strategies. A second cohort will have these same strategies applied utilizing the VDR/HFPV. Out come measures will include; ICU/Hospital length of stay, pulmonary infectious complications, airway pressure related complications, PaO2/PaCO2 levels, hemodynamic profiles, and ventilators days.

We hypothesize that patients with Acute Lung Injury (ALI )and/or Acute Respiratory Distress Syndrome (ARDS) managed primarily with HFPV will have fewer ventilators days, fewer infectious complications, and shorter ICU/hospital lengths of stay than patients managed with conventional mechanical ventilation techniques, while maintaining similar oxygenation (PaO2), ventilation (PaCO2), metabolic (pH), and hemodynamic (cardiac output) parameters.

ARDS and ALI have been shown to cause elevations in circulating inflammatory mediators as well as local (alveolar) mediators. The presence of increased amounts of both circulating and alveolar cytokines (inflammatory mediators) has been associated with increased mortality in patients with ARDS/ALI. The pulmonary capillary bed is a rich source of these inflammatory cytokines and the effects of ventilator strategies on circulating and compartmentalized (alveolar) cytokine levels may affect outcome.

Specific Aim 2: Circulating and alveolar inflammatory mediators (IL-6, IL-1-beta, IL-10, and TNF-alpha) will be measured, and activation of other markers of increased synthesis of inflammatory mediators (NF-kappa B and p38 map kinase) will be determined in isolated peripheral blood and alveolar leukocytes.

We hypothesize that patients with ALI/ARDS managed with HFPV will have lower levels of circulating and alveolar pro-inflammatory cytokines (IL-6, IL-1-beta and TNF-alpha) as well as less activation of NF-kappa B and p38 MAP kinase from peripheral blood and alveolar leukocytes.

ELIGIBILITY:
Inclusion Criteria:

* PaO2/FiO2 < 300 for less than 24 hours (Ratio of Partial pressure of oxygen to Fraction of inspired oxygen)

Exclusion Criteria:

* Documented Pneumonia,
* Documented Congestive Heart Failure,
* Immunosuppression,
* Enrolled in other interventional trial,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Ventilator Associated Pneumonia | 28 days

SECONDARY OUTCOMES:
Cytokine profiles | 96 hours
Length of stay | 28 dyas
Ventilator Days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Randall Friese, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States